CLINICAL TRIAL: NCT02955576
Title: Efficacy of Microneedle Patch on Topical Ointment Treatment of Psoriasis
Brief Title: Microneedle Patch for Psoriatic Plaques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VC16DISI0128
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Psoriasis; Administration, Topical
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Placebo Comparator): All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment only.
  Interventions: Other: Control
- Patch group (Active Comparator): All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment with patches.
  Interventions: Device: Patch
- Microneedle patch group (Experimental): All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment with microneedle HA patches.
  Interventions: Device: Microneedle HA patch

INTERVENTIONS:
Device: Microneedle HA patch — The microneedle HA patch were made of hyaluronic acid with microneedles which can enhance the drug permeation. All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment with microneedle HA patches.
  Microneedle HA patch (Therapass®, RMD-6.5A) was prepared at Raphas Co., Ltd. (Cheonan, South Korea).
  Daivobet® containing the active ingredients calcipotriol - betamethasone dipropionate was applied.
  Arms: Microneedle patch group
Device: Patch — The patch were made of hyaluronic acid with no microneedles to rule out the occlusion effect of microneedle HA patch. All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment with patches.
  Daivobet® containing the active ingredients calcipotriol - betamethasone dipropionate was applied.
  The hyaluronic acid patch was prepared at Raphas Co., Ltd. (Cheonan, South Korea) for this clinical trial, not for sale.
  Arms: Patch group
Other: Control — All lesions were treated with topical calcipotriol - betamethasone dipropionate ointment only.
  Daivobet® containing the active ingredients calcipotriol - betamethasone dipropionate was applied.
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy of microneedle patch on the psoriatic plaques.

DETAILED DESCRIPTION:
As a novel minimally invasive approach, microneedle-mediated transdermal drug delivery has received increased attention. Microneedle patch effectively penetrates the skin barrier of the stratum corneum and create efficient pathways for the delivery of drugs.

A randomized controlled trial based on split-body was planned to evaluate the efficacy of enhanced transdermal delivery of topical agent by hyaluronic acid (HA)-fabricated microneedle patch in psoriatic plaques. Six psoriatic plaques in a patient will be randomized to either microneedle HA patch, patch, or control groups. Patch group is planned for rule out the occlusion effect of patches. All lesions will be treated with topical agent and patches daily for 2-week period. The severity of psoriasis will be grated with modified PASI score and the clinical improvement will be assessed as % from baseline every week. Overall 20 patients with 120 psoriatic plaques will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 19
* A patient with psoriasis
* A patient with symmetrical psoriatic lesions
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages

Exclusion Criteria:

* Age: lower than 20
* A pregnant or lactating patient
* A patient who cannot understand the study or who does not sign the informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The improvement of psoriasis | Baseline, 1 week, 2 weeks
  The severity of psoriasis will be graded with modified PASI score, and the improvement will be assessed as % from baseline by using a computer program.

SECONDARY OUTCOMES:
The adverse effects of microneedle patch | Baseline, 1 week, 2 weeks
  It will be assessed by patient-report.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Min Bae, MD, PhD, Study Chair — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ju HJ, Kim JY, Jeong DH, Lee MS, Kim GM, Bae JM, Lee JH. Additional Use of Hyaluronic Acid-Based Dissolving Microneedle Patches to Treat Psoriatic Plaques: A Randomized Controlled Trial. Ann Dermatol. 2025 Apr;37(2):105-113. doi: 10.5021/ad.24.024. PMID 40165568